CLINICAL TRIAL: NCT01168063
Title: Medico-economic Evaluation of a Therapeutic Strategy Based on Molecular Detection of Antibiotic Resistance in the Management of H Pylori Infection
Brief Title: Molecular Detection of Antibiotic Resistance and H Pylori Eradication
Acronym: HELICOSTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P090210
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Diagnostic molecular testing; Antibiotic resistance; Treatment protocols
MeSH Terms: interventions — Quinolones; Clarithromycin; Metronidazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Helicobacter pilory triple treatment (Experimental): Triple treatment on this arm is based on results of molecular detection of resistance to antibiotics
  Interventions: Drug: Molecular detection of antibiotic resistance
- Helicobacter pilori standard recommended treatment (Active Comparator): H.Pylori Eradication rate with empirical treatment
  Interventions: Drug: standard triple therapy (PPI, amoxicillin, clarithromycin, metronidazole)

INTERVENTIONS:
Drug: Molecular detection of antibiotic resistance — Helico DR®, triple therapy (Proton Pomp Inhibitor (PPI), amoxicillin, clarithromycin, metronidazole)
  Other Names: Helicobacter Molecular detection of resistance to clarithromycin and quinolones; Use of triple therapy base on antibiotics resistances (PPI,amoxicillin,clarithromycin, metronidazole)
  Arms: Helicobacter pilory triple treatment
Drug: standard triple therapy (PPI, amoxicillin, clarithromycin, metronidazole) — 2 lines of treatments :
  1) PPI + Amoxicillin + Clarithromycin for 7 days
  1) PPI + Amoxicillin + Metronidazole for 14 days
  Other Names: Standard triple therapy (PPI, amoxicillin, clarithromycin, metronidazole ….)
  Arms: Helicobacter pilori standard recommended treatment

SUMMARY:
H pylori eradication failure with recommended triple therapy is mainly related to antibiotic resistance. However,IN VITRO culture of H pylori is uneasy and is not performed in routine practice. A molecular test of antibiotic resistance easy to perform is now available. The aim of the study was to compare eradication rates obtained with the standard treatment and with a treatment guided by the results of the molecular detection of antibiotic resistance.

DETAILED DESCRIPTION:
At the present time, H pylori infection is treated with a standard triple therapy. Treatment of naïve patients with triple therapy ( PPI+amoxicillin+clarithromycin for 7 days) markedly decreased last years to reach 70% due to a clarithromycin resistance rate about 20% in France. In case of failure, the recommended second line treatment (PPI+amoxicillin+metronidazole for 14 days) gives a success rate of 60%. However, as culture is uneasy and is only possible in specialised labs sensitivity to antibiotics is not currently studied before treatment.

The aim of the study was to evaluate clinical and medico-economic benefit of the molecular detection of antibiotic resistance in order to guide the treatment.

The test is performed after DNA extraction from biopsy specimens taken at gastroscopy allowing rapid detection of H pylori and clarithromycin or quinolone resistance.

Patients with bacteriologically proven H pylori infection will be randomly allocated to either empirical usual treatment with PPI , amoxicillin 1g, clarithromycin 500 mg X 2 /day for 7 days in naïve patients and PPI, amoxicillin 1g,metronidazole 500 mg X 2 /day for 14 days in patients who failed a first line treatment , or to treatment guided by the molecular test: PPI , amoxicillin 1g, clarithromycin 500 mg X 2 /day for 7 days in case of sensitivity to clarithromycin.In case of resistance to clarithromycin, quinolone should be given and in case of resistance to quinolone clarithromycin should be given. In case of resistance to both antibiotics metronidazole should be given.

Eradication will be assessed by performing 4 weeks after the completion of treatment with Urea Breath Test.

ELIGIBILITY:
Inclusion Criteria:

* H pylori infection bacteriologically confirmed
* Age > 18 years
* Naïve patient or one failure of the first line recommended treatment
* Patient referred to one out of the centres participating in the study

Exclusion Criteria:

* H pylori positive patient with at least failure of two lies of treatment
* patients with previous adverse event with PPI, amoxicillin, clarithromycin, levofloxacin or metronidazole
* PPI or antibiotic treatment in progressor stopped for less than 4 weeks
* patient with other severe sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate (at 3months according to the two strategies: empirical treatment versus treatment guided by molecular detection of antibiotic resistance) | at 3 months
  at 3 months according to the two strategies: empirical treatment versus treatment guided by molecular detection of antibiotic resistance

SECONDARY OUTCOMES:
Comparative cost of the two strategies | at 6 months according to the two strategies

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Delchier, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Result] Breuer T, Graham DY. Costs of diagnosis and treatment of Helicobacter pylori infection: when does choosing the treatment regimen based on susceptibility testing become cost effective? Am J Gastroenterol. 1999 Mar;94(3):725-9. doi: 10.1111/j.1572-0241.1999.00943.x. PMID 10086658
- [Derived] Delchier JC, Bastuji-Garin S, Raymond J, Megraud F, Amiot A, Cambau E, Burucoa C; HELICOSTIC Study Group. Efficacy of a tailored PCR-guided triple therapy in the treatment of Helicobacter pylori infection. Med Mal Infect. 2020 Sep;50(6):492-499. doi: 10.1016/j.medmal.2019.06.001. Epub 2019 Jun 27. PMID 31257067